CLINICAL TRIAL: NCT03197532
Title: Follicular and Luteal Dysfunction in Cancer Survivors
Brief Title: Assessing Urinary Hormones in Female Cancer Survivors
Acronym: AUHS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 811323
Record Dates: First submitted 2013-07-22; First posted 2017-06-23 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Effects of Chemotherapy
Keywords: fertility; hormones; healthy; chemotherapy; oncofertility; alkylating agent; fertility after cancer; late effects; survivorship; healthy volunteers; perimenopause; middle age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — daily urinary collections for 2 menstrual cycles
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Otherwise healthy, mid-reproductive aged women between the ages of 20 and 35 years previously exposed to high dose alkylating agent therapy (or have an alkylator score of 1 or more), and at least 1 year from cancer treatment.
- Group 2: Healthy, mid-reproductive aged women between the ages of 20 to 35 who have not been exposed to cancer therapy.
- Group 3: Reproductive aged women between the ages of 43-50 who have not been exposed to cancer therapy, nor have a history of infertility

SUMMARY:
Women of late to mid reproductive age may participate in a study using novel methodology to identify subtle changes in the reproductive endocrine axis via daily urine hormone analysis, which may have important implications for reproduction and may signal reproductive senescence.

DETAILED DESCRIPTION:
Women with a reduced follicular pool either from natural aging or previous chemotherapy, may not have any clinical signs or symptoms and traditional measures of ovarian reserve, such as basal Follicle Stimulating Hormone may be within the normal range. However, there may be alterations in the luteal or follicular phases(shortened follicular phase and luteal insufficiency) due to compromised follicle competency and alterations in the H-P-O axis. Therefore this aim uses novel methodology to identify subtle changes in the reproductive endocrine axis which may have important implications for reproduction and may signal reproductive senescence. Compared to yearly follicular measures of reproductive hormones, daily urine hormone analysis provides a more integrative assessment.

Three groups of subjects will be recruited:

Group 1: Otherwise healthy, mid-reproductive aged women between the ages of 20 and 35 years previously exposed to high dose alkylating agent therapy (or have an alkylator score of 1 or more), and at least 1 year from cancer treatment.

Group 2: healthy, mid-reproductive aged women between the ages of 20 to 35 who have not been exposed to cancer therapy.

Group 3: healthy, late reproductive aged women between the ages of 43-50 who have not been exposed to cancer therapy, nor have a history of infertility.

Subjects in all groups must have regular menstrual cycles every 21-35 days, and have a uterus and both ovaries. Each participant will complete daily urinary collections for 2 menstrual cycles to assess reproductive hormones. The ultimate goal of this work is to better estimate the reproductive window, or time to menopause.

ELIGIBILITY:
Inclusion Criteria for Group 1:

* Otherwise healthy, mid-reproductive aged women between the ages of 20 and 35 years previously exposed to high dose alkylating agent therapy (or have an alkylator score of 1 or more), and at least 1 year from cancer treatment.

Inclusion Criteria for Group 2:

* Healthy, mid-reproductive aged women between the ages of 20 to 35 who have not been exposed to cancer therapy.

Inclusion Criteria for Group 3:

* Healthy, late reproductive aged women between the ages of 43-50 who have not been exposed to cancer therapy, nor have a history of infertility.

Exclusion Criteria for all subjects:

* Pregnancy or lactation within the previous 3 months
* Use of hormonal contraception or replacement within the previous 3 months
* Body Mass Index greater than 30 kg/m2
* Excessive exercise greater than 1 hour per day
* Any medical condition other than cancer known to be associated with premature ovarian failure (such as Turners Syndrome or Fragile X) or ovulatory dysfunction (such as thyroid disease, congenital adrenal hyperplasia, Cushings syndrome, hyperprolactinemia, and polycystic ovary syndrome)

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Regularly menstruating postmenarchal, mid-reproductive aged female cancer patients treated with high dose alkylating agent chemotherapy or with an alkylator score of 1 or more.
  * Unexposed, regularly menstruating mid-reproductive aged women, and unexposed, regularly menstruating late reproductive aged women.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Urinary Follicle Stimulating Hormone (FSH) | up to 49 days each menstrual cycle
  Integrated urinary follicular-phase Follicle Stimulating Hormone (FSH) in urine samples collected daily for 2 menstrual cycles will be measured in mIU/mL by means of two-site chemiluminescent immunoassay with the use of two monoclonal antibodies.
Urinary Luteinizing Hormone (LH) | up to 49 days each menstrual cycle
  Integrated urinary follicular-phase Luteinizing Hormone (LH) in urine samples collected daily for 2 menstrual cycles will be measured in mIU/mL by means of two-site chemiluminescent immunoassay with the use of two monoclonal antibodies.
Urinary Estrone Conjugate (E1C) | up to 49 days each menstrual cycle
  Estrone Conjugate (E1C) in urine samples collected daily for 2 menstrual cycles will be measured in ug/dL by means of E1C immunoassay.
Urinary Pregnanediol-glucuronide | up to 49 days each menstrual cycle
  Pregnanediol-glucuronide (PDG) in urine samples collected daily for 2 menstrual cycles will be measured in ug/mL by means of PDG immunoassay.
Urinary Creatinine | up to 49 days each menstrual cycle
  Urinary Creatinine in urine samples collected daily for 2 menstrual cycles will be measured in mg/mL by means of spectrophotometric assay.

SECONDARY OUTCOMES:
Luteal and follicular phase lengths | up to 49 days each menstrual cycle
  Participants will be provided with calendars on which to record detailed menstrual cycle information during the study. The total menstrual cycle length will be defined as the number of days from day 1 of menses to the day before the next menses. The Kassam method will be used to determine evidence of luteal activity, presumably ovulation. Follicular phase will be defined as the number of days from day 1 of menses up to the day of luteal transition and the luteal phase length will be defined as the number of days beginning from the day after the day of luteal transition to the day before the next menses.

CONTACTS AND LOCATIONS:
Overall Officials: Clarisa R Gracia, MD, MSCE, Principal Investigator — University of Pennsylvania, Reproductive Research Unit
Locations (1):
- University of Pennsylvania, Reproductive Research Unit, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No